CLINICAL TRIAL: NCT00121290
Title: A Phase I Dose Escalation Study of Daily x 3 Intravenous SJG-136 in Patients With Advanced Solid Tumors
Brief Title: SJG-136 in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00085; NCI-2009-00085 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000653877; PHI 0453 (Other: Vanderbilt-Ingram Cancer Center); 6816 (Other: CTEP); P30CA068485 (NIH); U01CA099177 (NIH)
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 1,1'-((propane-1,3-diyl)dioxy)bis(7-methoxy-2-methylidene-1,2,3,10,11,11a-hexahydro-5H-pyrrolo(2,1-c)(1,4)benzodiazepin-5,11-dione)

ARMS (1):
- Treatment (SJG-136) (Experimental): Patients receive SJG-136 IV over 20 minutes once daily on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: SJG-136; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: SJG-136 — Given IV
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of SJG-136 in treating patients with solid tumors that are metastatic or cannot be removed by surgery. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of SJG-136 in patients with metastatic or unresectable solid tumors.

II. Determine the safety and dose-limiting toxic effects of this drug in these patients.

III. Determine, preliminarily, the efficacy of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetic parameters of this drug and its metabolites in these patients.

II. Correlate pharmacokinetic parameters with clinical effects of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive SJG-136 intravenously (IV) over 20 minutes once daily on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of SJG-136 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Prior chemotherapy or immunotherapy allowed
* Time interval must be at least 4 weeks since prior chemotherapy or immunotherapy, 6 weeks if the last regimen included BCNU or mitomycin C
* Radiation therapy to < 25% of hematopoietic bone marrow is allowed
* ECOG performance status =<2 (Karnofsky >= 60%)
* Life expectancy of greater than three months
* Recovered from prior therapy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine =< 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* No unstable angina pectoris

Exclusion Criteria:

* Patients receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SJG-136, breastfeeding should be discontinued if the mother is treated with SJG-136
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SJG-136
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with SJG-136
* With the exception of alopecia (and other situations in which the organ dysfunction or symptoms are considered clinically insignificant or irrelevant to this study), patients may not have baseline organ dysfunction or symptoms that qualify as Grade 2 or greater by CTC AE v. 3.0
* No other chemotherapy, immunotherapy, radiation therapy, surgery for cancer (including resection of any metastases), specific antitumor therapy, or experimental medications will be permitted while the patients are participating in this study
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Palliative radiation therapy is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-02; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity | 21 days

SECONDARY OUTCOMES:
Bivariate response variable (tumor response) evaluated by the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Igor Puzanov, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States